CLINICAL TRIAL: NCT04503564
Title: Feasibility of an Investigational Extended Wear Infusion Set for Continuous Subcutaneous Insulin Infusion (CSII) in Type 1 Diabetes Mellitus (T1DM) Participants
Brief Title: "FEXIS": (Feasibility of an Extended Wear CSII Set in Participants With T1DM)
Acronym: FEXIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capillary Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 150-1072-00; ACTRN12620000021976 (Registry Identifier: ANZCTR (Australian New Zealand Clinical Trials Registry)
Record Dates: First submitted 2020-07-09; First posted 2020-08-07 (Actual); Results first posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2022-05

CONDITIONS: Diabetes Mellitus, Type 1; Type 1 Diabetes; Type 1 Diabetes Mellitus; Diabetes Mellitus, Insulin-Dependent, 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: This study is designed as a single arm device feasibility evaluation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Achilles Infusion Set (Experimental): Coil-reinforced soft polymer indwelling cannula
  Interventions: Device: coil-reinforced soft polymer indwelling cannula

INTERVENTIONS:
Device: coil-reinforced soft polymer indwelling cannula — This is a prospective, non-randomized, home-use feasibility study of device performance, usability, tolerability, and safety of the Capillary Biomedical, Inc. (CapBio) Achilles infusion set for continuous subcutaneous insulin infusion (CSII or insulin pump therapy) in up to 20 participants diagnosed with type 1 diabetes mellitus (T1DM).

SUMMARY:
Over 1 million patients globally currently manage their Type 1 Diabetes mellitus using continuous subcutaneous insulin infusion with an infusion set that needs to be changed every 3 days. This study will assess the feasibility and device performance of the study device, the Achilles infusion set over three periods during routine insulin infusion.

This study will include 20 participants and has 3 periods:

Period 1 (up to 7 days): Trial run with study device with saline infusion. Period 2 (up to 7 days): participants will manage their blood glucose solely with their insulin pump and the Achilles infusion set. Blood glucose will be closely monitored with a continuous glucose monitoring (CGM) device.

Period 3 (up to 7 days): Participants will return to study center to receive a fresh Achilles infusion set and continue blood glucose management at home until infusion set failure or 7 days.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, home-use feasibility study of device performance, usability, tolerability, and safety of the Capillary Biomedical, Inc. (CapBio) Achilles infusion set for continuous subcutaneous insulin infusion (CSII or insulin pump therapy) in up to 20 participants diagnosed with type 1 diabetes mellitus (T1DM).

The CapBio Achilles infusion set is a sterile single use device designed to be used with commercially available infusion pumps (e.g., Medtronic MiniMed). The investigational Achilles infusion set contains a coil reinforced soft polymer indwelling cannula with one distal and three proximal holes.

The primary objective of this study is to determine feasibility and device performance of the CapBio Achilles infusion set over 2 extended home use wear periods of up to 7 days each during routine therapeutic insulin infusion. Feasibility is evidenced by the absence of uncontrolled hyperglycemia and/or suspected infusion set cannula occlusion.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is 18 - 70 years of age inclusive
2. Participant is in generally good health, as determined by the investigator
3. Participant is willing and able to individually complete written informed consent and agrees to comply with all study related testing and examinations
4. Participant must be geographically stable (e.g., expects to be available and capable of returning for all study specified test and examinations) during the study period
5. Participant has been diagnosed with T1DM for at least 12 months
6. C-peptide less than 0.6 nmol per L at screening
7. Subject can provide a minimum of 14 days of insulin pump data to demonstrate pump use compliance
8. Participant is willing to perform serum ketone measurements whenever the blood glucose is determined to be greater than 250 mg per dL (14 mmol per L) using a ketone meter and strips provided by the sponsor
9. Participant has BMI in the range 20 - 35 kg per square metre inclusive
10. Participant has experience infusing a rapid-acting insulin analog for at least 6 months
11. Participant has been using an insulin pump with commercially available infusion sets for at least 6 months (this includes Automated Insulin Delivery systems)
12. Participant has previous experience using a continuous glucose monitor (CGM) and is willing to use a CGM for the duration of the study and perform necessary calibration fingerstick glucose readings
13. Participant has ability to understand and comply with protocol procedures and to provide informed consent
14. AST and ALT less than or equal to 120 U per L
15. Creatinine less than 1.8 mg per dL

Exclusion Criteria:

1. Participants whose average total daily insulin dose exceeds 85 units per day (i.e. typically change insulin reservoirs more often than every 3.5 days on average)
2. Participants who routinely change their commercial insulin infusion sets twice weekly or less often (wear time greater than 3.5 days)
3. Female participant is pregnant or nursing (Documented negative pregnancy test results for female participants required unless participant is menopausal without any spontaneous menstrual cycles for >12 months or key organs have been removed.)
4. Participant has abnormal skin at intended device infusion sites (existing infection, inflammation, burns, or other extensive scarring)
5. Participant has HbA1C greater than 8.5 percent at screening
6. Participant has documented history in last 6 months of severe hypoglycemia associated with cognitive dysfunction sufficiently severe to require third party intervention or a history of impaired awareness of hypoglycemia.
7. Participant has a history of diabetic ketoacidosis in the last 6 months
8. Participant has known cardiovascular disease considered to be clinically relevant by the investigator
9. Participant has known arrhythmias considered to be clinically relevant by the investigator
10. Participant has known history of:

    1. Cushing's Disease,
    2. pancreatic islet cell tumor, or
    3. insulinoma
11. Participant has:

    1. Lipodystrophy,
    2. extensive lipohypertrophy, as assessed by the investigator
12. Participant is undergoing current treatment with:

    1. Systemic oral or intravenous corticosteroids,
    2. monoamine oxidase (MAO) inhibitors,
    3. non-selective beta-blockers,
    4. growth hormone,
    5. thyroid hormones, unless use has been stable during the past 3 months
13. Subject has significant history of any of the following, that in the opinion of the investigator would compromise the subject's safety or successful study participation:

    1. Alcoholism,
    2. drug abuse
14. Significant acute or chronic illness, that in the investigator's opinion, might interfere with subject safety or integrity of study results
15. Planned operation, MRI or CT which require removal of infusion set or CGM sensor during wear periods
16. Current participation in another clinical drug or device study
17. AST and ALT greater than 120 U per L
18. Creatinine equal to or greater than 1.8 mg per dL -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2020-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David O'Neal, M.D., Principal Investigator — St Vincent's Hospital Department of Medicine
Locations (1):
- St Vincent's Hospital (Melbourne) Ltd - Fitzroy, Melbourne, Australia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from existing participant population at study center. First patient was screened at medical clinic on 11/13/19
Pre-assignment Details: Screening period was up to 21 days. The study comprised of Week 1 with Achilles infusion set and saline and Weeks 2 and 3 with Achilles infusion set and insulin.
Groups:
- Achilles Infusion Set: Subjects used their own insulin infusion pumps from week 1 to 3. During week 1, participants wore 2 pumps. They wore their own pump (with insulin) and their own commercial infusion set and an additional study pump (with saline) and the investigational Achilles infusion set. During week 2-3, participants wore one pump. They wore their own pump (with insulin) and investigational Achilles infusion set.
Period: Achilles Infusion Set w/Saline- Week 1
Arm/Group | Achilles Infusion Set
Started | 20
Completed | 20
Not Completed | 0
Period: Achilles Infusion Set w/Insulin Week 2
Arm/Group | Achilles Infusion Set
Started | 20
Completed | 20
Not Completed | 0
Period: Achilles Infusion Set w/Insulin Week 3
Arm/Group | Achilles Infusion Set
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Achilles Infusion Set
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Median (Standard Deviation); unit: years] | 44.3 (14.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 1
BMI [Mean (Standard Deviation); unit: kg/m2] | 29.0 (4.01)

OUTCOME MEASURES:

1. Primary Outcome: Rate of Infusion Set Survival at End of Day 7
Description: The composite primary objective of this study is to evaluate feasibility and device performance of the Achilles infusion set over three extended home use wear periods of up to 7 days each during routine therapeutic insulin infusion.
Time Frame: 7 days during weeks 2 and 3
Population: Subjects used their own insulin infusion pumps from week 1 to 3. During week 1, participants wore 2 pumps. They wore their own pump (with insulin) and their own commercial infusion set and an additional study pump (with saline) and the investigational Achilles infusion set. During week 2-3, participants wore one pump. They wore their own pump (with insulin) and investigational Achilles infusion set.
Measure: Count of Units; unit: Achilles infusion sets
Units Other Than Participants: Achilles infusion sets
Arm/Group | Achilles Infusion Set
Number analyzed (Participants) | 20
Number analyzed (Achilles infusion sets) | 41
Achilles infusion sets | 36

ADVERSE EVENTS:
Time Frame: 3 weeks
Arm/Group | Achilles Infusion Set
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 15/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Achilles Infusion Set (N=20)
Dental caries (Gastrointestinal disorders) | 1 (1)
Dental Discomfort (Gastrointestinal disorders) | 1 (1)
Infusion site dryness (General disorders) | 1 (1)
Infusion site erythema (General disorders) | 5 (5)
Infusion site pain (General disorders) | 2 (2)
Infusion site pruritis (General disorders) | 1 (1)
Infusion site reaction (General disorders) | 1 (1)
Infusion site infection (Infections and infestations) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 7 (7)
Patient-Device Incompatibility (Product Issues) | 1 (1)
Skin lesion removal (Surgical and medical procedures) | 1 (1)
Separation Problem (General disorders) | 1 (1) — Infusion set got caught on door and pulled out

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-27): https://cdn.clinicaltrials.gov/large-docs/64/NCT04503564/Prot_SAP_000.pdf